CLINICAL TRIAL: NCT01732874
Title: Docosahexaenoic Acid Supplementation of Mothers to Improve Preterm Infant Nutrition and Immune Homeostasis
Brief Title: DHA Supplementation for Lactating Mothers
Acronym: DHA-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-0329
Record Dates: First submitted 2012-10-31; First posted 2012-11-26 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-10

CONDITIONS: Docosohexaenoic Acid Supplementation of Mothers to
Keywords: DHA; Preterm infant; Inflammation; Growth; Developement
MeSH Terms: conditions — Premature Birth; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expecta 200 mg (Other): Breastfeeding mothers of pre-mature infants randomly assigned to 200 mg Expecta to be taken orally once a day. Expecta to be taken for approximately 8 weeks post-partum or a shorter time if infant is discharged sooner from NICU.
  Interventions: Drug: Expecta 200 mg
- Expecta 1 Gram (Other): Breastfeeding mothers of pre-mature infants randomly assigned to one Gram of Expecta to be taken orally once a day. Expecta to be taken for approximately 8 weeks post-partum or a shorter time if infant is discharged sooner from NICU.
  Interventions: Drug: Expecta 1 gram

INTERVENTIONS:
Drug: Expecta 200 mg — Breastfeeding mothers who have given birth to premature infant 29 weeks or less will be randomized to receive 200mg Expecta. They will take once a day for 8 weeks or a shorter time if infant is discharged sooner from NICU.
  Other Names: Prenatal Dietary Supplement
  Arms: Expecta 200 mg
Drug: Expecta 1 gram — Breastfeeding mothers who have given birth to premature infant 29 weeks or less will be randomized to receive 1 gram of Expecta. They will take once a day for 8 weeks or a shorter time if infant is discharged sooner from NICU.
  Other Names: Prenatal Dietary Supplement
  Arms: Expecta 1 Gram

SUMMARY:
The purpose of this research study is to find out whether preterm infants are receiving enough of the essential and long chain fatty acids important for brain development and immune function. Our current intravenous (IV) fats do not contain the long chain fatty acids and different milk sources have different compositions. We would like to evaluate lactating mothers dietary intake and breastmilk level of fatty acid status by doing an analysis of their blood and breastmilk samples after they have been supplemented with a currently used fatty acid supplement (DHA- Martek Biosciences, now known as Dutch State Mines (DSM) Nutritional Lipid) The DHA supplement is available over the counter.

The information learned from this research study may benefit other mothers and babies in the future. The information could help make sure premature babies are receiving the right nutrients they need for appropriate growth and development.

DETAILED DESCRIPTION:
We designed a prospective, randomized trial to test the hypotheses that DHA supplementation to human milk providers will increase DHA concentration in milk and infant blood levels; and that infants receiving milk from DHA-supplemented providers will be receiving a more appropriate enteral intake to better mimic intrauterine accretion. In addition, we hypothesize that pro-inflammatory cytokines will be reduced in the mothers and infants receiving the higher DHA diet.

ELIGIBILITY:
Inclusion Criteria:

•Lactating mothers at Cincinnati University Hospital with infants born at < 29 weeks gestation.

Exclusion Criteria:

* the presence of congenital anomalies (trisomy 13, 18, 21, urethral, gastrointestinal and cardiac defects) that affect the standard course of care.
* mother's <18 and
* mothers with known allergy to algeal source
* mothers with history of bleeding disorders or taking any other medication that may increase the risk of bleeding
* infants with bleeding disorders or receiving any other medication that may increase the risk of bleeding

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ardythe Morrow, PhD, Principal Investigator — University of Cincinnati; Henry Akinbi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati University Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Valentine CJ, Dingess KA, Kleiman J, Morrow AL, Rogers LK. A Randomized Trial of Maternal Docosahexaenoic Acid Supplementation to Reduce Inflammation in Extremely Preterm Infants. J Pediatr Gastroenterol Nutr. 2019 Sep;69(3):388-392. doi: 10.1097/MPG.0000000000002375. PMID 31058771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers recruited at The University of Cincinnati with pregnancy < 28 weeks and no congenital anomalies
Period: Overall Study
Arm/Group | Expecta 200 mg | Expecta 1 Gram
Started | 16 | 11
Completed | 8 | 8
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Death of Infant | 3 | 2

BASELINE CHARACTERISTICS:
Population: Lactating mothers at Cincinnati University Hospital with infants born at < 29 weeks gestation admitted to The Cincinnati University Hospital NICU
Groups:
- Total: Total of all reporting groups
Arm/Group | Expecta 200 mg | Expecta 1 Gram | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 11 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 11 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Baseline Infant Serum Soluble Receptor for AGE (sRAGE) levels [Median (Inter-Quartile Range); unit: pg/ml] — sRAGE levels in infant serum samples at 0 weeks old from mothers supplemented with 200 or 1000 mg/kg per day of DHA. Serum Soluble Receptor for AGE (sRAGE) levels range from 7300-100 pg/mL where the higher number means a worse outcome.
  pg/ml | 746 [428 to 2201] | 5336 [416 to 7270] | 3041 [416 to 7270]

OUTCOME MEASURES:

1. Primary Outcome: Infant Serum Soluble Receptor for AGE (sRAGE) Levels at 4 Weeks From Baseline From Mothers Supplemented With 200 or 1000 mg/kg Per Day of DHA
Description: The study was powered to detect differences in sRAGE levels in infant serum samples at 4 weeks of age from mothers supplemented with 200 or 1000 mg/kg per day of DHA. Serum Soluble Receptor for AGE (sRAGE) levels range from 7300-100 pg/mL where the higher number means a worse outcome.
Time Frame: value at week 4
Population: Lactating mothers of pre-mature infants
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Expecta 200 mg | Expecta 1 Gram
Number analyzed (Participants) | 16 | 11
pg/mL | 900 [218 to 1650] | 1127 [256 to 2050]

ADVERSE EVENTS:
Time Frame: baseline to 4 weeks
Arm/Group | Expecta 200 mg | Expecta 1 Gram
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 0/16 | 0/11

LIMITATIONS AND CAVEATS:
The small sample size prevented the use of Repeated Measures Analyses, which would have given the study more power to detect differences and the ability to statistically control for any of the infant morbidities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT01732874/Prot_SAP_000.pdf